CLINICAL TRIAL: NCT00082550
Title: PET Imaging of Monoamine Transporters in OCD-related Disorders
Brief Title: Serotonin Transporters in Obsessive-Compulsive-Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040180; 04-M-0180
Record Dates: First submitted 2004-05-12; First posted 2004-05-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Genetics; Serotonin Transporter; Brain Imaging; Neurotransmitter; OCD; Obsessive-Compulsive Disorder; PET; Obsessive Compulsive Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Obsessive-Compulsive Disorder

SUMMARY:
This study will compare serotonin transporters in patients with obsessive-compulsive disorder (OCD) and healthy volunteers in order to better understand the role of serotonin in OCD. Serotonin is a chemical in the brain that transmits nerve impulses. The serotonin transporter (SERT) is a protein that regulates serotonin levels in the brain.

Normal, healthy volunteers and patients with OCD between 18 and 50 years of age and in overall good health may be eligible for this study. Candidates are screened with a medical history, physical examination, blood and urine tests, and a psychological interview and tests related to OCD symptoms. Participants undergo the following tests:

* Positron emission tomography (PET) scanning: For this test, subjects lie on the scanner bed, wearing special masks that are fitted to their heads and attached to the beds to help keep their heads still during the procedure. An 8-minute "transmission" scan is done to provide measures of the brain that will help calculate information obtained from subsequent scans. Then, a radioactive tracer is injected into a catheter (plastic tube) placed in the arm. The scan produces images of the serotonin transporters in the brain. Pictures are taken for about 2 hours, while the subject lies still on the scanner bed.
* Magnetic resonance imaging (MRI) scanning: An MRI scan of the brain is done within 1 year of the PET scan-that is, up to 1 year before or 1 year after the PET scan. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the patient lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 1 hour, during which the patient will be asked to lie still for up to a few minutes at a time.
* Genotyping: Subjects provide a blood sample (4 tablespoons) for DNA testing to look for genes or gene regions that may contribute to serotonin activity. This may lead to a better understanding of the genetic underpinnings of the serotonin system that influence mood, movement, and addiction.

DETAILED DESCRIPTION:
Evidence suggests that the symptoms of obsessive-compulsive disorder (OCD) arise from dysfunction of both the serotonergic and dopaminergic neurotransmitter systems. These two neurotransmitter systems are presumed to play a key modulatory role at the limbic-motor interface of the fronto-subcortical circuitry. However, in vivo knowledge linking the serotonergic and dopaminergic systems to OCD and OCD-related disorders is limited. In the current protocol, we plan to use PET to image the serotonin transporter (SERT) within the new radioligand [11C]DASB, in order to delineate regional abnormalities in SERT binding in drug-naive or drug-free OCD patients in comparison to healthy volunteers. In addition, we plan to examine the relationship between the regional PET measures of SERT and clinical severity measures of OCD. The goal of the present study is, thus, to further our understanding of the role of the serotonergic system in the pathophysiology of OCD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients and Controls:

Age: 18-65.

Patients- DSM-IV criteria for OCD.

Controls- not required

Patients and Controls:

Good health, with absence of serious medical illnesses, such as congestive heart failure, diabetes, kidney failure, epilepsy or cancer.

EXCLUSION CRITERIA:

Healthy Subjects:

History or current DSM-IV Axis I diagnostic criteria.

Patients and Controls:

Current diagnosis of major depressive disorder.

Patients and Controls:

Psychotropic medications, including SSRIs and antipsychotic medications. Drug free period must be greater than 4 weeks.

Patients and Controls:

Claustrophobia

Patients and Controls:

Pregnancy. Women with child bearing potential.

Patients and Controls:

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits.

Patients and Controls:

Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-05-10; Study Completion 2007-04-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bellodi L, Sciuto G, Diaferia G, Ronchi P, Smeraldi E. Psychiatric disorders in the families of patients with obsessive-compulsive disorder. Psychiatry Res. 1992 May;42(2):111-20. doi: 10.1016/0165-1781(92)90075-e. PMID 1631248